CLINICAL TRIAL: NCT03728218
Title: Visual Outcomes for Toric Efficacy Study
Acronym: VOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Kathryn Richdale, Associate Professor, University of Houston
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001070
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Astigmatism; Myopia
MeSH Terms: conditions — Astigmatism; Myopia | interventions — Contact Lenses

STUDY DESIGN:
Intervention Model Description: This is a crossover study of two types of contact lenses (toric orthokeratology and soft multifocals).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Orthokeratology Contact lenses (Experimental)
  Interventions: Device: Contact lenses (Orthokeratology)
- Soft Multifocal Contact lenses (Experimental)
  Interventions: Device: Contact lenses (Soft Multifocal)

INTERVENTIONS:
Device: Contact lenses (Orthokeratology) — Contact lenses
  Arms: Orthokeratology Contact lenses
Device: Contact lenses (Soft Multifocal) — Contact lenses
  Arms: Soft Multifocal Contact lenses

SUMMARY:
This is a crossover study of two types of contact lenses (toric orthokeratology and soft multifocals). Primary aims are to quantify correction of astigmatism, subjective and objective visual performance, aberrometry, peripheral refraction and bacterial bioburden between toric orthokeratology and soft toric multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 39 years of age (inclusive)
* Able to read and understand the study informed consent
* Plano to -5.00 D (inclusive) vertex corrected sphere power in each eye
* 1.25 to -3.50 D (inclusive) vertex corrected astigmatism in each eye
* Best corrected acuity of 20/25 or better in each eye
* No history of ocular pathology or surgery
* No significant binocular vision or accommodation abnormality (i.e. strabismus, amblyopia)
* No gas permeable lens wear for at least 1 month
* No systemic or ocular contraindications for contact lens wear
* Not pregnant/lactating (by self-report)

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Students for whom one of the principal investigators have direct access to/influence on grades would be consented and seen by another investigator for all visits.
* Pregnant/lactating women (by self-report)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Distance low contrast visual acuity | Up to two hours
  Monocular and binocular logMAR visual acuity

SECONDARY OUTCOMES:
Residual refractive error measured monocularly by cyclopleged auto-refraction | Up to two hours
  Cycloplegic auto-refraction to measure residual myopia/hyperopia and astigmatism

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

REFERENCES:
- [Background] Cheung SW, Cho P. Subjective and objective assessments of the effect of orthokeratology--a cross-sectional study. Curr Eye Res. 2004 Feb;28(2):121-7. doi: 10.1076/ceyr.28.2.121.26236. PMID 14972717
- [Background] Berntsen DA, Barr CD, Mutti DO, Zadnik K. Peripheral defocus and myopia progression in myopic children randomly assigned to wear single vision and progressive addition lenses. Invest Ophthalmol Vis Sci. 2013 Aug 27;54(8):5761-70. doi: 10.1167/iovs.13-11904. PMID 23838771
- [Background] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R, Suzaki A. The effects of entrance pupil centration and coma aberrations on myopic progression following orthokeratology. Clin Exp Optom. 2015 Nov;98(6):534-40. doi: 10.1111/cxo.12297. Epub 2015 Aug 17. PMID 26283026
- [Background] Benavente-Perez A, Nour A, Troilo D. Axial eye growth and refractive error development can be modified by exposing the peripheral retina to relative myopic or hyperopic defocus. Invest Ophthalmol Vis Sci. 2014 Sep 4;55(10):6765-73. doi: 10.1167/iovs.14-14524. PMID 25190657
- [Background] Kleinstein RN, Jones LA, Hullett S, Kwon S, Lee RJ, Friedman NE, Manny RE, Mutti DO, Yu JA, Zadnik K; Collaborative Longitudinal Evaluation of Ethnicity and Refractive Error Study Group. Refractive error and ethnicity in children. Arch Ophthalmol. 2003 Aug;121(8):1141-7. doi: 10.1001/archopht.121.8.1141. PMID 12912692
- [Background] Berntsen DA, Kramer CE. Peripheral defocus with spherical and multifocal soft contact lenses. Optom Vis Sci. 2013 Nov;90(11):1215-24. doi: 10.1097/OPX.0000000000000066. PMID 24076542
- [Background] Van Meter WS, Musch DC, Jacobs DS, Kaufman SC, Reinhart WJ, Udell IJ; American Academy of Ophthalmology. Safety of overnight orthokeratology for myopia: a report by the American Academy of Ophthalmology. Ophthalmology. 2008 Dec;115(12):2301-2313.e1. doi: 10.1016/j.ophtha.2008.06.034. Epub 2008 Sep 20. PMID 18804868
- [Background] Luo M, Ma S, Liang N. Clinical efficacy of toric orthokeratology in myopic adolescent with moderate to high astigmatism. Eye Sci. 2014 Dec;29(4):209-13, 218. PMID 26016072
- [Background] Chen C, Cheung SW, Cho P. Myopia control using toric orthokeratology (TO-SEE study). Invest Ophthalmol Vis Sci. 2013 Oct 3;54(10):6510-7. doi: 10.1167/iovs.13-12527. PMID 24003088
- [Background] Zimmerman AB, Nixon AD, Rueff EM. Contact lens associated microbial keratitis: practical considerations for the optometrist. Clin Optom (Auckl). 2016 Jan 29;8:1-12. doi: 10.2147/OPTO.S66424. eCollection 2016. PMID 30214344
- [Background] Bullimore MA, Sinnott LT, Jones-Jordan LA. The risk of microbial keratitis with overnight corneal reshaping lenses. Optom Vis Sci. 2013 Sep;90(9):937-44. doi: 10.1097/OPX.0b013e31829cac92. PMID 23892491
- [Derived] Tomiyama ES, Richdale K. Clinical Outcomes of a Randomized Trial with Contact Lenses for Astigmatic Myopia Management. Optom Vis Sci. 2023 Jan 1;100(1):9-16. doi: 10.1097/OPX.0000000000001969. Epub 2022 Dec 6. PMID 36705710
- [Derived] Tomiyama ES, Logan AK, Richdale K. Corneal Elevation, Power, and Astigmatism to Assess Toric Orthokeratology Lenses in Moderate-to-High Astigmats. Eye Contact Lens. 2021 Feb 1;47(2):86-90. doi: 10.1097/ICL.0000000000000721. PMID 32568927